July 30, 2013

Integrated Psychological Therapy (IPT) + Emotional Management Therapy (EMT) in chronic schizophrenia: study protocol for a randomized controlled trial





## **Osasun Mentaleko Sarea**

Red de Salud Mental

## Gipuzkoa

## **Information letter**

In San Sebastián, ......20

We hereby inform you that we are in a position to initiate the integrated psychological rehabilitation program for patients with chronic schizophrenia.

The program will consist of:

- Two evaluation sessions
- Eight months of psychological therapy, two sessions per week, one hour long.
- Evaluation sessions at the end of the program and follow-up at the month, three, six and twelve months.

The goal of the program is to achieve an improvement in symptoms, a better quality of life and a higher level of well-being.

The program will be applied in the Psychiatric Rehabilitation Unit of San Sebastián or in the reference health center.

We thank you for your interest in working with us, Best regards,

Program therapist: María Ruiz-Iriondo.

Study directors: Dr. Karmele Salaberria Irizar and Dr. Enrique Echeburúa.

All data obtained during the program are absolutely confidential, and will be used in accordance with what is established in Organic Law 15/1999, of December 13, on the protection of personal data.